CLINICAL TRIAL: NCT02191501
Title: Endoscopic Suturing of the Gastric Pylorus to Delay Gastric Emptying and Treat Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended as we are looking for more durable method/device
Sponsor: Northwell Health (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Larry Miller, PI, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Feinstein IRB#13-037B
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Over Weight
Keywords: Obesity Treatment; Endoscopy; Pyloric Suturing; Pyloric restriction
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyloric restriction (Experimental): Endoscopic method of pyloric restriction in order to decrease gastric emptying. The hypothesis is that this will cause and early and prolonged satiety which will inturn lead to decreased food consumption and lead to weight loss.
  Interventions: Procedure: Pyloric restriction

INTERVENTIONS:
Procedure: Pyloric restriction — The Apollo Overstitch Suturing Device is FDA approved for suturing in the gastrointestinal tract.
  However, the suturing device has never been used for suturing the pylorus in humans before. This procedure is not standard medical care. The safety and effectiveness of this procedure are being tested.

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of endoscopic suturing of the gastric pylorus to delay gastric emptying and treat obesity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, technical feasibility, and effectiveness of a endoscopic guided treatment for obesity - endoscopic pyloric suturing. The hypothesis and rationale for the study is that gastric pyloric restriction will cause early and prolonged satiety which will lead to decreased food intake and eventual weight loss. Both safety and efficacy of endoscopic pyloric suturing has been demonstrated in an animal model.

Screening of the participant is done 6-8 weeks prior to the procedure. Screening includes general history and physical examination, biochemical and laboratory analysis and informed consent. A baseline patient visit is performed 4-6 weeks prior to the procedure. The baseline visit involves a four hour gastric emptying scan in order to determine the rate of emptying of the stomach, the regional emptying of the upper and lower stomach, and the frequency and amplitude of contractions in the lower stomach. The baseline visit also includes nutritional counselling.

The procedure is performed in the endoscopy suite as an outpatient procedure. Patient will be prepped following usual practices and placed in a left lateral decubitus position. Following induction of sedation or anesthesia by the anesthesia provider, a complete endoscopic evaluation of the esophagus, stomach and jejunum following standard medical practices will be performed. The endoscope with mounted suturing device is advanced through an over-tube to the antrum and assess target area for stitch placement (physician will select appropriate target site in relation to participant's anatomy). The number of sutures required will vary for each procedure based on the size of the pylorus; however, it is thought that one or two sutures across the pylorus will be sufficient enough to achieve a functional restriction of the pylorus.

Participants will to be observed for a minimum of 1 hour following the procedure to monitor for adverse events. Patients will be recommended to take the following medications in order to minimize complications following pyloric suturing procedure; Proton Pump Inhibitor Omeprazole 40 mg recommended daily for 1 week prior to planned procedure date - and 40 mg twice daily after the procedure, Anti-Emetic -- Reglan or Zofran at the end of procedure and as needed after the procedure, and Scopalamine Patch to prevent nausea and vomiting.

All participants will be required to adhere to the follow-up schedule outlined below unless they have withdrawn their consent or died. The reason(s) the participant is not followed will be documented by the investigator. Follow-up for all participants will include a telephone contact at 1 and 18 weeks and clinic visits at 2,4, 8,10,12 and 24 weeks. At the 4 week visit, the participants will undergo a repeat four hour gastric emptying scan. At 3 months after the procedure participants will undergo repeat endoscopy to access the stomach and the suture site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65
* Male or female participants with a BMI >30 and < 45
* Female participants of childbearing age should not be pregnant, must have a negative serum or urine test and agree to use birth control for duration of the study.
* Participant did not undergo previous Roux-en-Y bypass with the gastric pouch limited to the cardia

Exclusion Criteria:

* Allergic to eggs or egg products, wheat, Gluten or Prolamins.
* currently on life saving oral medications
* Participants allergic to Scopolamine
* Participants allergic to botulinum toxin
* Participants who are currently on oral medications for their serious medical conditions.
* Recent tobacco cessation (within 3 months prior to planned enrollment) or plan to quit smoking during the study
* Infection anywhere in the body at time of procedure or other diseases that would make participant unsuitable for treatment (e.g., systemic disease, HIV, malignancy, autoimmune disease, etc.)
* patients who cannot undergo endoscopy
* Active disease of the gastrointestinal tract including esophageal inflammation, varices or ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis
* Esophageal or cricopharyngeal narrowing or stricture; distorted esophagus or known esophageal pouch
* Heavily scarred, malignant, or poor quality (e.g., friable or overly compliant) tissue in area to be sutured
* Severe eating disorders such as bulimia (use of purgatives/laxatives) or anorexia nervosa
* Significant movement limitations of lower extremities (e.g., cannot walk without the use of, or assistance from, a brace, cane, crutch, another person, prosthetic device, wheelchair, or other assistive device or is severely limited in their ability to walk due to an arthritic, neurological, or orthopedic condition)
* Recently (within previous 3 months) prescribed or initiated therapy with medication(s) known to cause significant weight gain or likely to require treatment with such medication(s) during the study OR is currently taking or has taken within the previous 3 months prescription or over-the-counter weight loss medications (e.g., medications and/or supplements containing ephedrine, phenylpropanolamine, amphetamines, etc.). Additionally, use of such medications and weight loss/appetite suppressing dietary supplements are prohibited during the course of the trial including the screening period
* Participant has history of significant cardiovascular or pulmonary disease (e.g., myocardial infarct, unstable angina, congestive heart failure, pulmonary edema or COPD) or other significant cerebrovascular disease (e.g., stroke)
* Not a candidate for general or conscious/moderate sedation
* Participant is on anticoagulant therapy (heparin, coumadin, Plavix, Ticlid, etc.) and must discontinue use of 325 mg aspirin within 6 weeks of procedure
* Active substance abuse (e.g., alcohol or drugs). This is done with personal interview only. No drug tests are being performed to determine the active abuse
* The participant has life expectancy of less than 1 year due to other medical conditions
* The participant is currently enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this trials study endpoints
* Patients having Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Percent weight loss | At 1, 3 and 6 months
  The primary endpoint of this study is percent weight loss at 1, 3 and 6 months (using the weight taken at the baseline visit as the baseline weight). Percent weight lost will be calculated as follows: [(Baseline Weight - Final 6 month Weight)/Baseline Weight] x 100%.

SECONDARY OUTCOMES:
Participant satisfaction | At 6 months post procedure
  Participant satisfaction with clinical outcomes at 6 months post-procedure will be captured on an ordinal scale of 1 to 5 with 1 representing very satisfied and 5 representing not satisfied at all. The response will be tabulated and presented using descriptive statistics.
Delay in gastric emptying | From baseline to 4 weeks post procedure
  A gastric emptying scan will be done prior to the endoscopic suturing procedure and four weeks after the endoscopic procedure to determine the rate of emptying of the stomach, the regional emptying of the upper and lower stomach, and the frequency and amplitude of contractions in the lower stomach.
Change in BMI | At 1, 3 and 6 Months
  BMI at 1, 3 and 6 months will be tabulated and summarized using descriptive statistics.
Percentage of Responders | At 1, 3 and 6 Months
  Percentage of participants losing at least 5%, 10%, 15% and 20% of weight at 1, 3 and 6 months will be tabulated and reported.
Change in Medication Use. | At 1, 3 and 6 Months
  If the participant is taking any medications for Obesity related complications such as Hypertension and Diabetes, then the dosage of those medications at 1, 3 and 6 months will be recorded and trends will be noted as either remained the same, decreased or increased.

CONTACTS AND LOCATIONS:
Overall Officials: Larry S Miller, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description and location of study — http://www.feinsteininstitute.org/clinical-research/clinical-research-studies/clinical-trial/13-037B/